CLINICAL TRIAL: NCT04387591
Title: Effect on Symptomatic Release of Remote Fu's Subcutaneous Needling on Patients With Biceps Tendinopathy
Brief Title: Fu's Subcutaneous Needling Treatment for Biceps Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Li-Wei Chou, Minister of Rehabilitation, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH107-REC3-026
Record Dates: First submitted 2020-05-10; First posted 2020-05-14 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Bicep Tendinitis
Keywords: Fu's Subcutaneous Needling; myofascial trigger point; muscle tone
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fu's subcutaneous needling(FSN) (Experimental): In this arm, the subjects will receive the intervention of FSN on Day1, Day2 and Day4, in total 3 treatments. The subjects will receive assessments before and after each interventions. After total treatments finished, the subjects will receive assessments on Day8 and Day15, separately.
  Interventions: Procedure: Fu's subcutaneous needling(FSN)
- Transcutaneous Electric Nerve Stimulation (Active Comparator): In this arm, the subjects will receive the intervention of Transcutaneous Electric Nerve Stimulation on Day1, Day2 and Day4, in the total 3 treatments. The subjects will receive assessments before and after each interventions. After total treatments finished, the subjects will receive assessments on Day8 and Day15, separately.
  Interventions: Procedure: Transcutaneous Electric Nerve Stimulation

INTERVENTIONS:
Procedure: Fu's subcutaneous needling(FSN) — In this study, the doctor will use a disposable Fu's subcutaneous needling(FSN) to penetrate the subject's skin of the middle of medial epicondyle and radial styloid process. Then the doctor will push forward the needle parallel to the skin surface (maintaining in the subcutaneous layer), towards the subject's medial epicondyle. The docotr will sway the needle 50 times in 30 seconds. After swaying the needle, the doctor will instruct the subject to do elbow flextion for 10 seconds resisting the doctor's opposite force, then the subject take a rest for 10 seconds. The above actions(elbow flexion and rest) are 3 repetitions. Then the subject do palmar flexion in the position of elbow flexion for 10 seconds resisting the doctor's opposite force, and take a rest for 10 seconds. These actions are also 3 repetitions. After the above reperfusion approach of muscles, the doctor will take out the needle to finish the treatment.
  Arms: Fu's subcutaneous needling(FSN)
Procedure: Transcutaneous Electric Nerve Stimulation — Transcutaneous electrical nerve stimulation (TENSor TNS) is the use of electric current produced bya device to stimulate the nerves for therapeuticpurposes. TENS, by definition, covers the completerange of transcutaneously applied currents usedfor nerve excitation although the term is often usedwith a more restrictive intent, namely to describe thekind of pulses produced by portable stimulators usedto treat pain. The unit is usually connected to theskin using two or more electrodes. A typical batteryoperated TENS unit is able to modulate pulse width,frequency and intensity. Generally TENS is applied athigh frequency (>50 Hz) with an intensity below motorcontraction (sensory intensity) or low frequency (<10Hz) with an intensity that produces motor contraction
  Arms: Transcutaneous Electric Nerve Stimulation

SUMMARY:
Biceps tendinopathy is a common cause in shoulder-pain symptoms. The major mechanism is overuse of the biceps muscles. The long-term accumulated and poor repaired trauma causes myofascial trigger points in the related muscles.We will conduct the randomized, open label experiment to evaluate the immediate, short-term, and long-term effect of Fu's subcutaneous needling (FSN).

DETAILED DESCRIPTION:
Biceps tendinopathy is a common cause in shoulder-pain symptoms. The major mechanism is overuse of the biceps muscles. The long-term accumulated and poor repaired trauma causes myofascial trigger points in the related muscles. Common symptoms are pain in the anterior shoulders and radiating pain in the biceps. Pain can be further elicited with lifting, pulling and repetitive overhead activity. Therefore, it can have a major impact on the patient's activity of daily life.

Fu's subcutaneous needling (FSN), as one of the dry needle treatments, performed by swaying a disposable Fu's subcutaneous needle parallel to the underlying muscles after penetrating the skin to the subcutaneous fascia. With the reperfusion activities, myofascial pain and soft tissue pain caused by myofascial trigger points can be decreased effective simultaneously. So far, there is no solid research or clinical trial to evaluate the efficacy of the treatment yet.

We will conduct the randomized, open label experiment to evaluate the immediate, short-term, and long-term effect of FSN. Outcome measures include visual analog scale, shoulder pain and disability index, pressure pain threshold, muscle tone changes and ultrasonographic evaluaton of biceps peritendinous effusion.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects older than 20 years of age who can cooperate with the experimental volunteers.
2. Suffering from biceps tendon lesions for more than one month, and subjective pain intensity (VAS) greater than 5 points.
3. There is a local tender point in front of the shoulder, and the shoulder joint pronation test can induce pain.
4. Under soft tissue ultrasound, the thickness of biceps peritendinous effusion (BPE) on the affected side of the biceps tendon is greater than1 mm.

Exclusion Criteria:

1. There are contraindications to general treatment, such as serious medical problems, recent serious trauma, or pregnant women.
2. There has been a history of drug abuse (including excess alcohol) that affects pain assessors.
3. Have received shoulder, neck or upper back surgery.
4. People with central or peripheral nerve disease.
5. Cognitive impairment, unable to cooperate with the experimenter.
6. Patients currently receiving other treatments for biceps tendinopathy.
7. Patients receiving shoulder injection treatments within the last 6 months.
8. Patients with rheumatic diseases.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scales | before and after Day1, Day2, Day4 treatment ; on Day8 and Day15 separately
  The visual analogue scale or visual analog scale is a psychometric response scale which can be used in questionnaires. This tool used to help a person rate the intensity of certain sensations and feelings, such as pain. A straight line of 100mm is actually marked with 0 mm on the far left and 100mm on the far right. Two faces are drawn on both ends. Explain to the patient that 0 mm means no pain and 100 mm means very painful. From the left end, the right shift indicates more and more pain. The evaluator will let the patient draw a short line vertically on the line,representing his painful position, and record the measured cm value. In this test, if the score of the subject decreases,it can represent the treatment is helpful for the improvement of the patient's pain.

SECONDARY OUTCOMES:
Pressure Pain Threshold | before and after Day1, Day2, Day4 treatment ; on Day8 and Day15 separately
  Pressure pain threshold (PPT) is defined as the minimum force applied which induces pain. This measure has proven to be commonly useful in evaluating tenderness symptom.
Muscle tension | before and after Day1, Day2, Day4 treatment ; on Day8 and Day 15 separately
  Muscle tension is the muscle's resistance to passive stretch during resting state. The measuring tool called Myotone will calculate three parameters such as tone, elasticity and stiffness and get a value to represent the muscle tension. If the value decrease, it can represent the treatment is helpful for the subjective muscle relax.
Shoulder pain and disability index (SPADI) | before and after Day1, Day2, Day4 treatment ; on Day8 and Day15 separately
  The Shoulder Pain and Disability Index (SPADI) is a patient-reported outcome measure. All question items in the survey are presented on a 10cm visual analog scale (VAS). The verbal anchors for the pain dimension are "no pain at all" and "worst pain imaginable." And the verbal anchors for the functional activities are "no difficulty" and "so difficult it requires help". The scores from both dimensions are averaged to derive a total score with 0 being the best outcome (less disability) and 100 the worst (greater disability). If the value decrease, it can represent the treatment is helpful for shoulder pain relief and functional activities.
Ultrasonographic evaluaton of biceps peritendinous effusion | before and after Day1, Day2, Day4 treatment ; on Day8 and Day15 separately
  The biceps tendon is evaluated in the bicipital groove with the arm in a neutral position and the hand resting palm up on the patient's thigh. If the biceps peritendinous effusion decrease, it can represent the treatment is helpful.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Wei Chou, PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided